CLINICAL TRIAL: NCT01031693
Title: Pilot Study of Transcranial Magnetic Stimulation (TMS) in Nicotine Addiction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Maryland (Other)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 999909440; 09-DA-N440
Record Dates: First submitted 2009-12-11; First posted 2009-12-14 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2013-08-28

CONDITIONS: Nicotine Dependence
Keywords: Nicotine; Cigarettes; Tobacco; Transcranial Magnetic Stimulation (TMS); Cue-Induced Craving; Smoking
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Transcranial Magnetic Stimulation

ARMS (2):
- Group A (Active Comparator): Active TMS
  Interventions: Device: Transcranial Magnetic Stimulation
- Group B (Sham Comparator): Sham TMS
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — daily sessions for 5 days

SUMMARY:
Background:

* Treatment for nicotine addiction is characterized by high rates of relapse. New treatment therapies for nicotine addiction are exploring the use of brain scanning equipment to control and decrease nicotine and cigarette cravings.
* Transcranial magnetic stimulation (TMS) uses magnetic pulses to stimulate the brain. These pulses can change activity in parts of the brain. Researchers are interested in determining whether TMS delivered in single pulses can decrease activity in the parts of the brain that respond to nicotine craving.

Objectives:

- To determine whether single pulse TMS can reduce cue-induced nicotine craving and use in cigarette smokers.

Eligibility:

* Individuals 18 years of age and older who are physically healthy and have smoked 10 or more cigarettes per day for at least 1 year.
* A small group of healthy nonsmoking control subjects 18 years of age and older will also participate in the study.

Design:

* The study will involve seven study visits and two follow-up visits. The control participants will have only two visits: one with a magnetic resonance imaging (MRI) scan and one with TMS to evaluate brain function and response.
* Participants will have an initial assessment about tobacco use habits and craving patterns, and will provide blood and urine samples before beginning the study.
* Participants will have two initial MRI brain scans. The first scan will look at the structure of the brain at rest. During the other scan, participants will look at images related to and not related to cigarette smoking.
* The single pulse TMS sessions (with either actual TMS or inactive [sham] TMS) will be held daily for 5 consecutive days. Magnetic pulses will be triggered by cigarette-related picture cues and delivered at varying intervals before the participant sees a cigarette-related picture. During these testing visits, researchers will ask questions related to tobacco use and craving, and collect urine and breath samples for further study.
* Participants will have two follow-up visits, 1 week and 2 weeks after the TMS sessions, to evaluate memory and mood, and will have one final MRI brain scan at the end of the study.

DETAILED DESCRIPTION:
Primary objective: Transcranial magnetic stimulation (TMS) provides a non-invasive means of inhibiting brain neural activity. This pilot study will test whether 5 days of single pulse (sp) TMS reduces cue-induced nicotine craving and use in cigarette smokers.

Hypothesis: We predict that active spTMS will significantly lower craving for nicotine compared with sham spTMS.

Study population: Subjects will be up to 73 adult cigarette smokers (averaging greater than or equal to 10 cigarettes daily for greater than or equal to one year) with current nicotine dependence (based on DSM-IV criteria or Faerstrom Test for Nicotine Dependence score greater than or equal to 3). Subjects will not have other current major psychiatric disorders or substance abuse. Subjects in the pilot phase (one fMRI and one TMS session to valid brain mapping procedures) will be up to 25 healthy non-smokers.

Design: Following a baseline day to evaluate subject characteristics, subjects will be randomly assigned to receive 5 days of active or sham spTMS session. spTMS at strength 120 percent of the motor threshold will be applied to the prefrontal cortex (PFC) using a figure-eight coil. Magnetic pulses will be triggered by cigarette-related pictorial cues and delivered at varying intervals prior to presentation of a cigarette-related picture. TMS pulses will not be delivered during emotionally salient images unrelated to nicotine or emotionally neutral images. Brain site localization will use a computerized navigation system based on functional and structural MRI scans obtained before the first session. Each session (lasting around 20 minutes) will consist of 108 trials (cue presentations): 72 with nicotine-associated cues and 18 each with non-drug-associated positive or neutral cues. Subjects return for follow-up fMRI and behavioral assessments one and two weeks after the final TMS session.

Outcome measures: The primary outcome measure will be nicotine craving assessed with the Tobacco Craving Questionnaire and visual analog scales before and after every TMS session and at one- and two-week follow-up. Secondary outcome measures will include cigarette smoking over the test period and at follow-up assessed by self-report, salivary cotinine levels, and expired breath CO levels. A follow-up fMRI will evaluate changes in regional brain activity associated with changes in craving and TMS treatments.

Benefits: Participants will not directly benefit from this study. This study may contribute to better scientific understanding of nicotine addiction and development of better treatment methods.

Risks: The primary risks from TMS are transient headache, scalp discomfort, and hearing loss (minimized by wearing ear plugs). Seizures are very rare when spTMS is administered within accepted safety guidelines and individuals at increased risk of seizures are excluded. By excluding individuals with a history of non-drug-induced mania/ hypomania we minimize the risk of inducing a manic episode.

ELIGIBILITY:
-INCLUSION CRITERIA:

i) Eighteen years of age or older

ii) Current nicotine dependence (by DSM-IV criteria or Fagerstrom Test for Nicotine Dependence score greater than or equal to 3) and averaging smoking 10 or more cigarettes per day for at least one year.

iii) Reading level of at least 6th grade, based on the Wide Range Achievement Test (WRAT)

iv) Ability to give valid informed consent

v) Right-handed

vi) If the subject is female, of childbearing potential, and sexually active, she agrees to use a medically acceptable contraception, and not become pregnant for the duration of the study. A woman is considered of childbearing potential unless post-menopausal or surgically sterilized. Female patients of childbearing potential who are or who anticipate the possibility of becoming sexually active with a male partner must use either: (1) contraceptive pill or IUD or depot hormonal preparation (ring, injection implant); and/or (2) a barrier method of contraception such as diaphragm, sponge with spermicide, or condom. Women who are not sexually active do not have to agree to use one of the acceptable contraception methods. Contraceptive measures will be reviewed with female subjects at each visit prior to the TMS session.

vii) Self-report experiencing nicotine craving when exposed to nicotine-associated cues

EXCLUSION CRITERIA:

i) Personal or first-degree family history of any clinically defined neurological disorder, including organic brain disease, epilepsy, stroke, brain lesions, multiple sclerosis, previous neurosurgery, or personal history of head trauma that resulted in loss of consciousness.

ii) Cardiac pacemakers, neural stimulators, implantable defibrillator, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease, with intracranial implants (e.g. aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head that cannot be safely removed.

iii) Metal shrapnel or bullet in the head or body including metal shavings.

iv) Current use of any investigational drug or of any medications with anti or pro-convulsive action

v) Increased intracranial pressure (lowers seizure threshold)

vi) Lifetime history of major depressive disorder, schizophrenia, bipolar disorder, mania, or hypomania

vii) History of myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, or any heart condition currently under medical care.

viii) Pregnant or nursing women or women with reproductive potential who are sexually active and not using an acceptable form of contraception.

ix) Any history of seizure

x) Current dependence (DSM-IV criteria) on substances other than nicotine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2009-07-13; Primary Completion 2013-08-28 (Actual); Study Completion 2013-08-28 (Actual)

PRIMARY OUTCOMES:
Nicotine craving by Tobacco Craving Questionnaire and visual-analogue scales. | 2 weeks

SECONDARY OUTCOMES:
Cigarette use by self-report, salivary cotinine level, and expired breath CO levels. | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David A Gorelick, M.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (2):
- United States (2):
  - National Institute on Drug Abuse, Baltimore, Maryland
  - Maryland Psychiatric Research Center (MPRC) 55 Wade Avenue, Catonsville, Maryland

REFERENCES:
- [Background] Allen EA, Pasley BN, Duong T, Freeman RD. Transcranial magnetic stimulation elicits coupled neural and hemodynamic consequences. Science. 2007 Sep 28;317(5846):1918-21. doi: 10.1126/science.1146426. PMID 17901333
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Bestmann S, Baudewig J, Siebner HR, Rothwell JC, Frahm J. Functional MRI of the immediate impact of transcranial magnetic stimulation on cortical and subcortical motor circuits. Eur J Neurosci. 2004 Apr;19(7):1950-62. doi: 10.1111/j.1460-9568.2004.03277.x. PMID 15078569